CLINICAL TRIAL: NCT00948909
Title: A Randomized, Double-Blind, Placebo- and Active-Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of ABT-126 in Subjects With Mild-to-Moderate Alzheimer's Disease
Brief Title: Efficacy and Safety Study for Subjects With Mild-to-Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M10-984; 2009-011424-64 (EudraCT Number)
Record Dates: First submitted 2009-07-24; First posted 2009-07-29 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Sugars; ABT-126; Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (4):
- A. Sugar Pill (Placebo Comparator)
  Interventions: Drug: Placebo
- B. ABT-126 (Experimental)
  Interventions: Drug: ABT-126
- C. ABT-126 (Experimental)
  Interventions: Drug: ABT-126
- D. donepezil (Active Comparator)
  Interventions: Drug: donepezil

INTERVENTIONS:
Drug: Placebo — Placebo intervention
  Other Names: Sugar Pill
  Arms: A. Sugar Pill
Drug: ABT-126 — Experimental intervention
  Arms: B. ABT-126; C. ABT-126
Drug: donepezil — Active comparator intervention
  Other Names: Aricept
  Arms: D. donepezil

SUMMARY:
This is a efficacy and safety study evaluating new treatment for subjects with mild to moderate Alzheimer's Disease.

DETAILED DESCRIPTION:
This is a Phase 2 study designed to evaluate the efficacy and safety of ABT-126 in approximately 260 adults with mild-to-moderate Alzheimer's disease (AD). Subjects will be randomized to one of the four treatment groups (ABT-126, donepezil, or placebo) for a 12-week Treatment Period. Acronyms are listed in the secondary outcome section, below, you will find a list of the acronyms defined:

* MMSE - Mini Mental Status Exam
* QoL-AD - Quality of Life - Alzheimer's Disease
* CIBIC-plus - Clinician Interview-Based Impression of Change
* NPI - Neuropsychiatric Inventory
* CSDD - The Cornell Scale for depression in Dementia
* ADCS-ADL - Alzheimer's Disease Cooperative Study - Activities of Daily Living

ELIGIBILITY:
Inclusion Criteria:

* The subject is a male or female between the ages of 55 and 90 years, inclusive, at Screening Visit 1.
* The subject meets the NINCDS/ADRDA criteria for probable AD.
* The subject has a Mini-Mental Status Examination (MMSE) total score of 10 to 24, inclusive, at Screening Visit 1.
* The subject has a Modified Hachinski Ischemic Scale (MHIS) score of less than or equal to 4 at Screening Visit 1.
* If female, subject must be postmenopausal for at least two years or surgically sterile
* The subject has an identified, reliable, caregiver.

Exclusion Criteria:

* The subject is currently taking or has taken a medication for the treatment of Alzheimer's disease or dementia within 60 days prior to Screening Visit 1
* The subject has a history of any significant neurologic disease other than AD.
* In the opinion of the investigator, the subject has any clinically significant uncontrolled medical or psychiatric illness.
* The subject has reported history of discontinuation of donepezil due to lack of efficacy.
* The subject has a history of intolerance or adverse reaction to donepezil that led to discontinuation.
* The subject has a known hypersensitivity to donepezil, piperidine derivatives, or any of the excipients in either donepezil hydrochloride or ABT-126 formulations.
* Patient uses non-prescribed drugs of abuse or has a history of drug or alcohol abuse/dependence.
* Subjects with AST and ALT values at Screening Visit 1 that are greater than or equal to 1.5-fold the upper limit of normal (ULN).

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2009-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
ADAS-Cog - Alzheimer's Disease Assessment Scale Cognition portion | Measurements up through 12 weeks.

SECONDARY OUTCOMES:
MMSE, QoL-AD, CIBIC-plus, NPI, CSDD, ADAS-Cog (13 item) and ADCS-ADL. Note: Acronyms are fully defined in the area titled Detailed Description. | Measurements up through 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Gault, MD, Study Director — AbbVie
Locations (29):
- United States (3):
  - Site Reference ID/Investigator# 19904, Fresno, California
  - Site Reference ID/Investigator# 23025, West Palm Beach, Florida
  - Site Reference ID/Investigator# 19905, Indianapolis, Indiana
- Bulgaria (4):
  - Site Reference ID/Investigator# 22944, Pleven
  - Site Reference ID/Investigator# 22942, Plovdiv
  - Site Reference ID/Investigator# 22945, Sofia
  - Site Reference ID/Investigator# 22946, Sofia
- Czechia (5):
  - Site Reference ID/Investigator# 20276, Litoměřice
  - Site Reference ID/Investigator# 20273, Pilsen
  - Site Reference ID/Investigator# 20274, Prague
  - Site Reference ID/Investigator# 20272, Prague
  - Site Reference ID/Investigator# 20701, Prague
- Slovakia (4):
  - Site Reference ID/Investigator# 23625, Bratislava
  - Site Reference ID/Investigator# 23624, Bratislava
  - Site Reference ID/Investigator# 23622, Michalovce
  - Site Reference ID/Investigator# 23942, Rimavská Sobota
- South Africa (7):
  - Site Reference ID/Investigator# 20267, Belville
  - Site Reference ID/Investigator# 20266, Cape Town
  - Site Reference ID/Investigator# 20261, Durban
  - Site Reference ID/Investigator# 21682, George
  - Site Reference ID/Investigator# 20265, Johannesburg
  - Site Reference ID/Investigator# 20271, Port Elizabeth
  - Site Reference ID/Investigator# 20263, Richards Bay
- United Kingdom (6):
  - Site Reference ID/Investigator# 20187, Blackburn
  - Site Reference ID/Investigator# 20183, Bradford
  - Site Reference ID/Investigator# 20191, Crowborough
  - Site Reference ID/Investigator# 20184, Glasgow
  - Site Reference ID/Investigator# 20190, London
  - Site Reference ID/Investigator# 20192, Southampton

REFERENCES:
- [Derived] Gault LM, Ritchie CW, Robieson WZ, Pritchett Y, Othman AA, Lenz RA. A phase 2 randomized, controlled trial of the alpha7 agonist ABT-126 in mild-to-moderate Alzheimer's dementia. Alzheimers Dement (N Y). 2015 Jun 23;1(1):81-90. doi: 10.1016/j.trci.2015.06.001. eCollection 2015 Jun. PMID 29854928